CLINICAL TRIAL: NCT01756274
Title: Performance of Three Bayer Blood Glucose Monitoring Systems With Blood Samples From Neonates
Brief Title: Evaluation of Blood Glucose Monitoring Systems With Blood Samples From Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2010-009-03
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neonates 'Left-over' Blood Samples (Experimental): Blood samples used in this study were 'left-over samples'. The blood samples were from heel sticks of neonates, collected (into a tube) and sent to the laboratory. Two left-over samples could be obtained from a single neonate. Laboratory professionals tested the BG concentration using three Bayer Blood Glucose Monitoring Systems (BGMS): Contour® NEXT BGMS, Contour® PLUS BGMS, and Contour® Next EZ BGMS.
  Interventions: Device: Contour® NEXT BGMS; Device: Contour® PLUS BGMS; Device: Contour® Next EZ BGMS

INTERVENTIONS:
Device: Contour® NEXT BGMS — Lab professionals tested the BG concentration using Contour® NEXT BGMS (Blood Glucose Monitoring System). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method, Cobas® 6000 instrument (Roche Diagnostics Corp., Indianapolis, IN).
Device: Contour® PLUS BGMS — Lab professionals tested the BG concentration using Contour® PLUS BGMS (Blood Glucose Monitoring System). All meter BG results were compared with capillary plasma results obtained with a reference laboratory glucose method, Cobas® 6000 instrument (Roche Diagnostics Corp., Indianapolis, IN).
Device: Contour® Next EZ BGMS — Lab professionals tested the BG concentration using Contour® Next EZ BGMS (Blood Glucose Monitoring System). All meter BG results were compared with plasma results obtained with a reference laboratory glucose method, Cobas® 6000 instrument (Roche Diagnostics Corp., Indianapolis, IN).

SUMMARY:
The purpose of this study was to evaluate the performance of three Bayer Blood Glucose Monitoring Systems (BGMS) with neonatal blood. Blood samples used in this study were 'left-over samples'. The blood samples were from heel sticks of neonates, collected (into a tube) and sent to the laboratory. All meter Blood Glucose (BG) results were compared with capillary plasma results obtained with a reference laboratory glucose method (Cobas® 6000 instrument).

ELIGIBILITY:
Inclusion Criteria:

* Routine blood samples (heelstick) collected from neonates (less than 30 days of age).
* A portion of the samples (approximately 10%) will be from subjects <24 hours old.
* A portion of the samples (at least 10%) will be from subjects in the NICU.
* Sample blood volume must be sufficient to complete investigational testing in addition to prescribed testing.

Exclusion Criteria:

* Samples from babies >=30 days of age

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J Dietzen, PhD, DABCC, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neonates 'Left-over' Blood Samples: Blood samples used in this study are 'left-over samples' from heel sticks of neonates, collected (into a tube) and sent to the laboratory. Lab professionals tested the BG concentration using 3 Bayer Blood Glucose Monitoring Systems: Contour® NEXT, Contour® PLUS, and Contour® Next EZ BGMS.
Period: Overall Study
Arm/Group | Neonates 'Left-over' Blood Samples
Started | 162
Completed | 159
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Laboratory error | 1

BASELINE CHARACTERISTICS:
Population: Of 217 blood samples from 162 neonates 211(217-6) were included in data analysis. Two samples could not be used because they had been taken from sources that had not been specified in the protocol. Four samples had no reference method results due to laboratory errors.
Units Other Than Participants: blood samples
Groups:
- Neonates 'Left-over' Blood Samples: Blood samples used in this study are 'left-over samples' from heel sticks of neonates, collected (into a tube) and sent to the laboratory. Lab professionals tested the BG concentration using 3 Bayer Blood Glucose Monitoring Systems: Contour® NEXT, Contour® PLUS, and Contour® Next EZ BGMS. Each subject could contribute up to 2 blood samples. Baseline Characteristics for Participant Flow based on number of blood samples, not number of subjects.
Arm/Group | Neonates 'Left-over' Blood Samples
Number analyzed (Participants) | 162
Number analyzed (blood samples) | 211
Age, Customized [Number; unit: blood samples]
  < 24 hours | 25
  1-29 days | 186
Sex/Gender, Customized [Number; unit: blood samples]
  Female | 100
  Male | 111
Region of Enrollment [Number; unit: blood samples]
  United States | 211
Nursery Location [Number; unit: blood samples]
  Special Care | 101
  Well Baby | 58
  NICU (Neonatal Intensive Care Unit) | 30
  Other | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent of Blood Glucose Results Within +/-15 mg/dL(<75 mg/dL) and Within +/-20% (>=75 mg/dL) of the Reference Instrument BG Value
Description: Laboratory professionals tested the BG concentration of 'left-over samples' using plasma referenced Blood Glucose Monitoring Systems. BGMS results were compared with capillary plasma BG results obtained with a Cobas® 6000 instrument (Roche Diagnostics Corp., Indianapolis, IN).
Time Frame: 30 minutes
Population: Each subject could contribute up to 2 blood samples. Of 217 blood samples 211(217-6) were included in data analysis. Two samples could not be used because they had been taken from sources that had not been specified in the protocol. Four samples had no reference method results due to laboratory errors.
Measure: Number; unit: percentage of Blood Glucose Results
Units Other Than Participants: Blood Samples
Groups:
- Neonates 'Left-over' Blood Samples: Blood samples used in this study were 'left-over samples' from heel sticks of neonates, collected (into a tube) and sent to the laboratory. Lab professionals tested the BG concentration using 3 Bayer Blood Glucose Monitoring Systems: Contour® NEXT, Contour® PLUS, and Contour® Next EZ BGMS. Each subject could contribute up to 2 blood samples.
Arm/Group | Neonates 'Left-over' Blood Samples
Number analyzed (Participants) | 159
Number analyzed (Blood Samples) | 211
percentage of Blood Glucose Results
  Contour® NEXT BGMS | 100.0
  Contour® PLUS BGMS | 99.5
  Contour® Next EZ BGMS | 99.5

2. Secondary Outcome: Percent of BG Results (Per Population) Within +/-15 mg/dL (<100 mg/dL)and Within +/-15% (>=100 mg/dL) of the Reference Instrument BG Value
Description: as for outcome 1
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Number; unit: percentage of BLOOD GLUCOSE RESULTS
Units Other Than Participants: BLOOD SAMPLES
Groups:
- Neonates 'Left-over' Blood Samples: Blood samples used in this study were'left-over samples' from heel sticks of neonates, collected (into a tube) and sent to the laboratory. Lab professionals tested the BG concentration using 3 Bayer Blood Glucose Monitoring Systems: Contour® NEXT, Contour® PLUS, and Contour® Next EZ BGMS. Each subject could contribute up to 2 blood samples.
Arm/Group | Neonates 'Left-over' Blood Samples
Number analyzed (Participants) | 159
Number analyzed (BLOOD SAMPLES) | 211
percentage of BLOOD GLUCOSE RESULTS
  Contour® NEXT BGMS | 99.5
  Contour® PLUS BGMS | 99.1
  Contour® Next EZ BGMS | 99.1

3. Other Pre Specified Outcome: Number of Blood Samples From Babies Less Than 24 Hours Old That Produced Meter Results Beyond What Random Chance Would Predict (i.e. Outside 95% Limits for Studentized Residuals)
Description: To evaluate the effect of neonatal age on the meter systems' performances, the number of blood samples that produced unusual meter results out of the total number of blood samples that came from babies less than 24 hours old was reported. Studentized residuals were used to measure the degree to which meter BG results departed from what would be expected using a linear model. (This analysis is not related to BGM accuracy status, which has already been reported.)
Time Frame: 30 minutes
Population: Of 217 'left-over' blood samples, 211(217-6) were included in data analysis. Of these, twenty five (25) blood samples were obtained from babies that were less than 24 hours old.
Measure: Number; unit: BLOOD SAMPLES
Units Other Than Participants: BLOOD SAMPLES From Babies <24 hours old
Arm/Group | Neonates 'Left-over' Blood Samples
Number analyzed (Participants) | 25
Number analyzed (BLOOD SAMPLES From Babies <24 hours old) | 25
BLOOD SAMPLES
  Contour® NEXT | 1
  Contour® PLUS | 2
  Contour® Next EZ | 1

4. Other Pre Specified Outcome: Number of Blood Samples From Babies in the Neonatal Intensive Care Unit (NICU) That Produced Meter Results Beyond What Random Chance Would Predict (i.e., Outside 95% Limits for Studentized Residuals)
Description: To evaluate how the meter systems perform with blood samples drawn in the Neonatal Intensive Care Unit, the number of blood samples that produced unusual meter results out of the total number of blood samples that came from babies in Neonatal Intensive Care was reported. Studentized residuals were used to measure the degree to which meter BG results departed from what would be expected using a linear model. (This analysis is not related to BGM accuracy status, which has already been reported.)
Time Frame: 30 minutes
Population: Of 217 'left-over' blood samples, 211(217-6) were included in data analysis and, of these, thirty (30) blood samples were obtained from babies in the Neonatal Intensive Care Unit (NICU).
Measure: Number; unit: BLOOD SAMPLES
Units Other Than Participants: BLOOD SAMPLES From Babies in the NICU
Arm/Group | Neonates 'Left-over' Blood Samples
Number analyzed (Participants) | 30
Number analyzed (BLOOD SAMPLES From Babies in the NICU) | 30
BLOOD SAMPLES
  Contour® NEXT | 4
  Contour® PLUS | 2
  Contour® Next EZ | 3

ADVERSE EVENTS:
Groups:
- Neonates 'Left-over' Blood Samples: Blood samples used in this study are 'left-over samples' from heel sticks of neonates, collected (into a tube) and sent to the laboratory.
Arm/Group | Neonates 'Left-over' Blood Samples
Serious Adverse Events (participants affected / at risk) | 0/162
Other Adverse Events (participants affected / at risk) | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days